CLINICAL TRIAL: NCT01003938
Title: Continuous Infusion Topotecan With Erlotinib for Topotecan Pretreated Ovarian Cancer: Tumor Features and Phase II/Pharmacokinetic Evaluation
Brief Title: Topotecan With Erlotinib for Topotecan Pretreated Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to administrative issue and financial sponsor decision to suspend ovarian cancer studies
Sponsor: NYU Langone Health (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYU 08-613
Record Dates: First submitted 2009-10-27; First posted 2009-10-29 (Estimated); Results first posted 2014-01-16 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-05

CONDITIONS: Ovarian Cancer
Keywords: chemotherapy; combination therapy; targeted therapy; second-line
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Topotecan; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- topotecan and erlotinib (Experimental): Topotecan 0.4 mg/m^2/day administered via continuous infusion for 9 days beginning on Day 1, every 21 days cycle; erlotinib 150 mg daily for 9 days every 21 days cycle. Both drugs will be given for a minimum of 2 cycles.
  Interventions: Drug: Topotecan; Drug: Erlotinib

INTERVENTIONS:
Drug: Topotecan
  Other Names: Topotecan hydrochloride; Hycamtin
Drug: Erlotinib
  Other Names: Tarceva

SUMMARY:
This is a single arm phase II study with a combination of Hycamptin® (topotecan) and erlotinib for a minimum of 2 cycles in patients (18 yrs of age and older) with recurrent ovarian cancer previously treated with chemotherapy drug Hycamptin® (topotecan). Up to 30 patients will be enrolled in this study.

DETAILED DESCRIPTION:
On Day 1 of each treatment cycle, topotecan 0.4 mg/m^2/day will be administered via continuous infusion for 9 days beginning on Day 1 of every 21 day cycle. Additionally, patients will receive erlotinib 150 mg daily Days 1-9 in a cycle of 21 days. Thereafter both drugs will be given as long as patient benefit continues. Treatment will be administered on an inpatient or outpatient basis, repeating administration on an every 3 week cycle.

A cycle will be one three-week course of the erlotinib-topotecan regimen (the cycle could be extended to 4 weeks if blood studies at 21 days result in treatment delay).

The dose of topotecan will be calculated as follows:

BSA (m^2) X drug dose (mg/m^2) = dose (mg)

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven, previously treated, epithelial ovarian cancer, and/or serous ovarian cancer.
2. Evaluable disease with CA125 levels two times the upper limit of normal for the institution (>50u/ml ) on two occasions at least one week apart is required in order to apply CA-125 response criteria.
3. Previously treated for ovarian cancer with a taxane and platinum based regimen. and an additional topotecan regimen (any number of chemotherapy or biologic therapies are allowed; including prior erlotinib are allowed)
4. Age >= 18 years.
5. Minimum life expectancy: 4 months.
6. ECOG (Eastern Cooperative Oncology Group) performance status 0,1, or 2. 0: Fully active, unrestricted activities of daily living. 1: Ambulatory, but restricted in strenuous activity. 2: Ambulatory, and capable of self care. Unable to work. Out of bed for greater than 50% of waking hours.
7. Complete blood count (CBC) performed less than seven days prior to enrollment and have an absolute neutrophil count >1.0 X 10^9/L, and a platelet count >100 X 10^9/L.
8. Serum chemistry panel drawn less than seven days prior to enrollment and have a total bilirubin <= 1.5 X the institutional upper limit of normal (IULN), or SGOT/AST is < 2.5 X IULN.
9. Serum creatinine <= 1.5 X institutional upper limit of normal (IULN). If the serum creatinine level is >= 1.5 IULN, but the serum creatinine clearance >= 50 mg/dL, then the subject can enter the study.
10. Central line access.
11. Signed written informed consent (approved by the Institutional Review Board [IRB]/Ethics Committee) obtained prior to study entry.

Exclusion Criteria:

If the answer to any of the exclusion criteria is YES, the subject is NOT ELIGIBLE for the study.

1. Presence of active cancer other than that described in Section 3.1.criteria (a), with the exception of a diagnosis of synchronous occurrence of adenocarcinoma in ovary and uterus.
2. Uncontrolled intercurrent illness not limited to infection, symptomatic congestive heart failure, or unstable angina pectoris, or cardiac arrhythmia.
3. Acute toxicity of prior chemotherapy is still present
4. History of severe allergic reaction to erlotinib
5. Unresolved sequelae resulting from any surgical procedures.
6. Symptomatic, untreated brain metastases. Patients with untreated brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
7. Lactating or pregnant. The investigational agent topotecan may be toxic to the developing fetus or nursing infant and poses unknown health risks. Documentation of a negative, serum HCG pregnancy test is required for women of child bearing potential (WOCBP) within 2 weeks prior to the start of treatment. WOCBP is defined as women who have not been naturally postmenopausal for at least 12 consecutive months or no previous surgical sterilization. A negative pregnancy test within 2 weeks prior to start of treatment is required.
8. Women of childbearing potential must use effective contraception throughout the time they are on study. Before entering this trial, patients must be made aware of the risk in becoming pregnant.
9. Receipt of any investigational drug within 28 days before beginning treatment with study drug and/or concomitant treatment with other investigational agents.
10. Patients with a history of poorly controlled gastrointestinal disorders that could affect absorption of erlotinib (e.g. Crohn's, ulcerative colitis, etc)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-08; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco Muggia, MD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - Bellevue Hospital Center, New York, New York
  - NYU Clinical Cancer Center, New York, New York
  - Tisch Hospital, New York, New York

REFERENCES:
- [Derived] Warner E, Liebes L, Levinson B, Downey A, Tiersten A, Muggia F. Continuous-infusion topotecan and erlotinib: a study in topotecan-pretreated ovarian cancer assessing shed collagen epitopes as a marker of invasiveness. Oncologist. 2014 Mar;19(3):250. doi: 10.1634/theoncologist.2013-0398. Epub 2014 Feb 21. PMID 24563078

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From Oct 2009 to May 2011, 6 patients were enrolled to this trial from New York University Medical Center and its affiliated hospitals.
Groups:
- Topotecan and Erlotinib: On Day 1 of each treatment cycle, topotecan 0.4 mg/m^2/day was administered via continuous infusion for 9 days beginning on Day 1, every 21 days cycle. Plus erlotinib 150 mg daily for 9 days every 21 days cycle.
Period: Overall Study
Arm/Group | Topotecan and Erlotinib
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Topotecan and Erlotinib
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 65 [61 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Prior regimens [Number; unit: participants]
  4 regimens | 1
  5 regimens | 3
  7 regimens | 1
  8 regimens | 1

OUTCOME MEASURES:

1. Primary Outcome: CA125 Response Rate With Continuous-infusion Topotecan and Erlotinib
Description: Response was assessed after every treatment cycle. Response rate is defined as number of the patients who experienced complete or partial CA125 response (CR or PR). CR: normalization of the CA125 value, determined by 2 observations not less than 4 weeks apart; PR: CA125 decreases by >50% and is confirmed to be 50% or greater on a subsequent determination at least one month later.
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | Topotecan and Erlotinib
Number analyzed (Participants) | 6
participants | 1

2. Secondary Outcome: CA125 Response Duration
Description: Response duration is measured from the time measurement criteria for CA125 CR/PR at the first met until the first date that recurrent or progressive disease is objectively documented.
Time Frame: Up to 3 years
Population: The study was terminated very early (6 enrolled vs. 30 target accrual). No statistical analysis was performed on patient data.
Arm/Group | Topotecan and Erlotinib
Number analyzed (Participants) | 0

3. Secondary Outcome: CA125 Stable Disease Duration
Description: Stable disease (SD) duration is measured from the tile of start of therapy until the criteria for progression are met. SD: CA125 decreases <50% or increases <100%. Disease progression: CA125 doubles the value of baseline, or more, over time.
Time Frame: Up to 3 years
Population: as for outcome 2
Arm/Group | Topotecan and Erlotinib
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Progression
Description: Time to progression is defined as the time from first study drug administration until the first day radiological and /or symptomatic disease progression is documented, or until death in the absence of progression.
Time Frame: Up to 3 years
Population: as for outcome 2
Arm/Group | Topotecan and Erlotinib
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: estimated total time from the start of the trial
Time Frame: 4 years
Population: as for outcome 2
Arm/Group | Topotecan and Erlotinib
Number analyzed (Participants) | 0

6. Secondary Outcome: Toxicity Profile
Description: Number of participants (patients) who experienced AEs.
  Dry skin, dry eye, acne, erythema, rash, pruritus, and diarrhea were related erlotinib; dehydration, anemia, leukopenia, nausea, vomiting, platelets, and fatigue were realted to topotcan.
Time Frame: the whole treatment phase and 30 days post-treatment
Measure: Number; unit: participants
Arm/Group | Topotecan and Erlotinib
Number analyzed (Participants) | 6
participants
  Dry skin (grade 1) | 2
  Dry skin (grade 3) | 1
  Dry eye (grade 1) | 1
  Acne (grade 1) | 2
  Erythema (grade 1) | 1
  Rash/ desquamation (grade 1) | 1
  Rash/ desquamation (grade 2) | 1
  Pruritis (grade 1) | 1
  Diarrhea (grade 1) | 2
  Diarrhea (grade 2) | 1
  Dehydration (grade 3) | 1
  Anemia (grade 2) | 2
  Anemia (grade 3) | 2
  Leukopenia (grade 2) | 3
  Leukopenia (grade 3) | 1
  Nausea (grade 1) | 4
  Nausea (grade 2) | 1
  Nausea (grade 3) | 1
  Vomiting (grade 1) | 3
  Vomiting (grade 2) | 1
  Vomiting (grade 3) | 1
  Platelets (grade 1) | 2
  Platelets (grade 2) | 1
  Platelets (grade 3) | 1
  Fatigue (grade 1) | 2
  Fatigue (grade 2) | 1
  Fatigue (grade 3) | 1

ADVERSE EVENTS:
Description: All adverse events are reported regardless of relationship to the therapy.
Arm/Group | Topotecan and Erlotinib
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topotecan and Erlotinib (N=6)
Dehydration (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topotecan and Erlotinib (N=6)
Anorexia (Gastrointestinal disorders) | 3
Ascites (non-malignant) (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
"Constitutional Symptoms-Other" (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
"Dermatology/Skin-Other" (Skin and subcutaneous tissue disorders) | 2
Diarrhea patients without colostomy (Gastrointestinal disorders) | 3
Dry eye (Eye disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dyspepsia/heartburn (Gastrointestinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
Dysuria (painful urination) (Renal and urinary disorders) | 1
Edema (Vascular disorders) | 1
"Fatigue (lethargy, malaise, asthenia)" (General disorders) | 4
Flatulence (Gastrointestinal disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 5
"Hemorrhage-Other (Specify, nosebleeds)" (Respiratory, thoracic and mediastinal disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Leukocytes (total WBC) (Investigations) | 4
Lymphopenia (Investigations) | 2
"Musculoskeletal-Other" (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2
"Pain-Other" (General disorders) | 2
Platelets (Investigations) | 4
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3
"Renal/Genitourinary-Other (Specify, urinary frequency)" (Renal and urinary disorders) | 1
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Weight loss (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes